CLINICAL TRIAL: NCT03510169
Title: Novel Use of Negative Pressure Assist in Neonates With Respiratory Distress: a Feasibility Study Using Neovest
Brief Title: Use of Gentle Synchronized Negative Pressure in Helping Babies Breathe
Acronym: Neovest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-282Neovest
Record Dates: First submitted 2018-04-05; First posted 2018-04-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Distress Syndrome; TTN; RDS of Prematurity; Respiratory Distress, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Distress Syndrome In Premature Infants; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoVest (Experimental): Negative pressure ventilation using NeoVest
  Interventions: Device: NeoVest

INTERVENTIONS:
Device: NeoVest — Negative pressure ventilation with NeoVest
  Other Names: Negative Pressure Ventilation

SUMMARY:
The NeoVest delivery device is a wearable vest/shell that surrounds the infant's abdomen. It was developed using serial body measurements of infants previously admitted to the St. Michael's Hospital NICU (REB #15-183). It gently pulls on the abdomen by applying negative pressure, thereby displacing the diaphragm. The materials used for the NeoVest are lightweight and suitable for the infants' sensitive skin.

The AIM of the present study is to demonstrate the feasibility of applying negative pressure NIV, that is synchronized and proportional to the infant's respiratory demand. The preliminary data on feasibility can be used to apply for larger grants from the CIHR, for a study of the NeoVest in smaller premature infants.

DETAILED DESCRIPTION:
Respiratory distress is a common reason why newborn infants require intensive care soon after birth. Premature infants are at risk of having immature lungs and/or weak respiratory muscles requiring the provision of respiratory support with a mechanical ventilator. Full term infants can also require respiratory support for lung disease or lung immaturity. The most commonly used form of non-invasive respiratory support is positive pressure delivered via nasal prongs or a nasal mask, also known as nasal continuous positive airway pressure (nCPAP). Nasal CPAP is thought to be effective in a variety of newborn lung disorders including respiratory distress syndrome, transient tachypnea of the newborn, etc. Although many forms of nCPAP exist, they are not typically synchronized to a baby's breathing efforts (1,2).

Furthermore, due to the infants' sensitive skin and underdeveloped nasal bridges, continued use of nasal devices can lead to skin breakdown and permanent damage to the nose (3). In order to provide optimal ventilation, these devices must be tight-fitting nasal interfaces to provide a leak-free environment (3). There is also variability in the success of nasal interfaces in providing uniform ventilation. This is because the positive pressure provided at the level of the infants' nostrils is dissipated (through the open mouth, etc.) as it travels down the infants' airways to the alveoli of their lungs (3). Additionally, prolonged use of nasal ventilation methods may impede infant bonding with their mothers via decreased skin-to-skin time, etc. Nasal CPAP is often cited as a reason why feeding (including breastfeeding) is delayed in babies requiring neonatal intensive care stay.

Negative pressure ventilation (NPV) involves the application of sub-atmospheric pressures around the abdomen to displace the diaphragm. It is a unique alternative for administering NIV to infants and would avoid complications associated with nasal interfaces. NPV has previously been used in treating infants with respiratory distress using old-fashioned, large and bulky "iron-lung" devices (4-12). One of the earliest studies using NPV for infants with respiratory failure showed that in a series of 26 patients, NPV provided a sustained increase in PaO2 (5). The infants were a mean gestational age of 32 to 33 weeks and met the criteria for respiratory failure defined by PaO2 < 40mmHg on 100% inspired oxygen and/or PCO2 > 70mmHg during bag-mask ventilation (5). Further studies on NPV, continued to show effectiveness in the ventilation of infants with lung disease with improved oxygenation (6-12).

In this study, the investigators propose a novel negative pressure interface and device that is synchronized to the infant's respiratory drive and provides intermittent application of negative pressure. The device utilizes Neurally Adjusted Ventilator Assist (NAVA) technology to achieve synchronization to the infant's underlying respiratory drive and control.

The electrical activity of the diaphragm (Edi) is measured using a specialized feeding tube catheter with miniaturized sensors at the end. There is a small balloon at the tip of the catheter that measures the gastric pressure which provides evidence that the diaphragm is being displaced. The Edi catheter has been shown in previous work to be effective in delivering both invasive and non-invasive positive pressure ventilation with the FDA-approved NAVA and a variety of interfaces (13-15). The Edi catheter is used routinely in many NICUs worldwide as a conventional nasal or oral catheter.

NAVA is a mode of ventilation that is neurally integrated with the inherent lung protective reflexes by utilizing the information obtained from the Edi catheter. During spontaneous breathing, as lung inflation progresses, stretch receptors in the lungs will eventually sense an adequate inspired volume, and "switch off" inspiration. For a patient on NAVA, where the neural inspiration also controls the assist delivery, the ventilator breath will be cycled-off when neural exhalation begins. Several studies have demonstrated that infants spontaneously choose lower peak inspiratory pressures (PIP) and tidal volume during NAVA compared to conventional ventilation (targeted by the clinician) (16-23).

"Traditional" NAVA is triggered on and off with the Edi and delivers assist proportionally to the Edi on inspiration only. The PEEP is fixed and defined by the clinician. During this "traditional NAVA" there is a fair amount of tonic Edi that is not assisted. With continuous NAVA, the Edi is used to continuously adjust the assist. The Edi controls both the inspiratory and expiratory assist. A safety and tolerance study in 20 preterm infants using neutrally adjusted PEEP (neuroPAP) was done using nasal prongs as the delivery interface (See Appendix 2).

In this study, the investigators plan to control a negative pressure delivery device (NeoVest) to deliver synchronized negative NIV for a short period of time. Preliminary data in small rats (~400g) and larger rabbits (~3-4kg) have demonstrated feasibility and efficacy in experimental conditions mimicking neonatal respiratory distress (See Appendix 3). The Neovest was able to generate multiple effective levels of ventilator support in these animals with no side effects.

The NeoVest delivery device is a wearable vest/shell that surrounds the infant's abdomen. It was developed using serial body measurements of infants previously admitted to the St. Michael's Hospital NICU (REB #15-183). It gently pulls on the abdomen by applying negative pressure, thereby displacing the diaphragm. The materials used for the NeoVest are lightweight and suitable for the infants' sensitive skin.

The AIM of the present study is to demonstrate the feasibility of applying negative pressure NIV, that is synchronized and proportional to the infant's respiratory demand. The preliminary data on feasibility can be used to apply for larger grants from the CIHR, for a study of the NeoVest in smaller premature infants.

ELIGIBILITY:
Inclusion Criteria:

* 20 infants, admitted to Neonatal Intensive Care Unit (NICU) at St. Michael's Hospital
* >1.5kg birthweight
* Clinically stable, with symptoms of respiratory distress (due to transient tachypnea of the newborn, respiratory distress syndrome, etc.)
* Stable on nasal CPAP (5-8cm H2O) for a minimum of 6 hours
* Within the first two weeks of life

Exclusion Criteria:

* Infants with FiO2 requirements >0.35
* Infants with clinically significant apnoea or bradycardia (> 2 A&B in last hour, or apnea >20 sec, or bradycardia requiring significant stimulation)
* Infants with hemodynamic instability (mean BP < weeks GA), or any infant requiring fluid boluses and/or inotropic medications
* Infants with genetic conditions or dysmorphic facial features
* Infants that have been recently extubated in the last 48 hours
* Infants in whom placement of the NG tube is contra-indicated
* Infants with any clinical suspicion of upper airway distress such as symptoms of stridor
* Infants with abdominal wall defects and other visible abnormalities of the abdomen or chest
* Infants with umbilical arterial and/or venous catheters
* Infants that have allergies and/or previous skin reactions to silicone based materials

Ages: 6 Hours to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of negative pressure ventilation with NeoVest | 22 minutes
  Ability to provide negative pressure ventilation with the NeoVest

SECONDARY OUTCOMES:
Diaphragm Electrical Activity | Will be obtained every 1-5 minutes, or following any change in respiratory support
  Obtained from Edi catheter
Respiratory Rate | Will be obtained every 1-5 minutes, or following any change in respiratory support
  Breaths per minute
Heart Rate | Will be obtained every 1-5 minutes, or following any change in respiratory support
  Beats per minute
Oxygen Saturation | Will be obtained every 1-5 minutes, or following any change in respiratory support
  Percent oxygen saturation
Transcutaneous Carbon Dioxide Level | Will be obtained every 1-5 minutes, or following any change in respiratory support
  Transcutaneous meassurement in mmHg
Blood Pressure | Will be obtained every 1-5 minutes, or following any change in respiratory support
  Obtained with blood pressure cuff in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Campbell, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital NICU, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No